CLINICAL TRIAL: NCT05453019
Title: Effects of Cochlear Implantation on Tinnitus and Its Symptoms
Brief Title: Effects of CI on Tinnitus and Its Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, YangShiming, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI and Tinnitus 01
Record Dates: First submitted 2022-06-22; First posted 2022-07-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Tinnitus
Keywords: tinnitus; electrical stimulation; cochlear implant
MeSH Terms: conditions — Tinnitus | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tinnitus group (Experimental): Patients who have tinnitus got cochlear implant
  Interventions: Device: Cochlear Implant
- without tinnitus group (Active Comparator): Patients who have no tinnitus got cochlear implant
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — The surgeon will make a small cut (incision) behind patient's ear, and form a small hole in the portion of skull bone (mastoid) where the internal device rests. Then the surgeon create a small opening in the cochlea in order to thread the electrode of the internal cochlear implant device. The skin incision is stitched closed so that the internal device is under the skin.

SUMMARY:
Abnormal activity in the central auditory system is the cause of subjective experience of tinnitus. Electrical stimulation can inhibit the abnormal activity of auditory related neurons in patients with tinnitus. In recent years, the application of electrical stimulation in the treatment of tinnitus is a hot research topic, and has made some progress. However, its treatment is still in the discussion stage, and there is no best scheme suitable for clinical practice. At present, scholars have found that cochlear electrode stimulation can inhibit tinnitus, but its mechanism is not clear. It is difficult to locate the origin of tinnitus, and the location of electrode stimulation and stimulation parameters still need to be further optimized. Because the implanted part of the cochlear implant contains magnets, the patients cannot perform functional MRI. However, the prevalence of tinnitus in this group is very high (67.0~100.0%, with an average of 80.0%), so it is of great value and significance to study the effect of tinnitus treatment in such patients. In this study, a new clinical electroencephalogram (EEG) technique was used to make up for the lack of MRI imaging in patients with electrode implantation. EEG analyzes the functional connection of different brain regions through EEG test electrodes, uses the traceability function of EEG software to locate the location of tinnitus, analyzes the process of tinnitus inhibition by electrical stimulation, and explains the mechanism of tinnitus inhibition by electrical stimulation from a new perspective.

DETAILED DESCRIPTION:
1. Research content 1.1 Study on the change law of tinnitus affected by electrical stimulation after electrode implantation: 1) The change of tinnitus before operation after cochlear implantation; 2) Long term observation of electrical stimulation after cochlear implantation: (1) The change rule of tinnitus loudness after electrical stimulation (how long can it recover to be stable after power on); (2) The regularity of tinnitus frequency after electrical stimulation; (3) The recovery of tinnitus after electrode implantation for various causes of deafness.

   1.2 Study on the mechanism of electric stimulation inhibiting tinnitus: 1) Changes of resting EEG in patients with tinnitus before surgery, before surgery-after surgery, 1 month, 2 months, 3 months, 6 months, 12 month, more than 12 months; 2) The compilation of resting electroencephalogram analysis program; 3) The resting brain wave shape was analyzed to trace the anatomical position of the artificial cochlea to inhibit tinnitus.

   1.3 Study on the optimal setting of electrode stimulation for tinnitus treatment: 1) Setting different electric stimulation frequency and stimulation rate parameters to mask tinnitus; 2) Set the procedure of electric stimulation cochlear implant to mask tinnitus.
2. Research objectives 1) Summarize the changes of tinnitus after electrode implantation (effective treatment time, diseases suitable for electrical stimulation treatment, etc.); 2) Infer the mechanism of electric stimulation inhibiting tinnitus; 3) Set electrical stimulation parameters to effectively suppress tinnitus.
3. Scientific problems to be solved Our study group plan to use more advanced EEG technology to explore the principle of electric stimulation to suppress tinnitus, find out the effective scheme of electric stimulation to treat tinnitus, and help more patients solve the problem of tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* 1. This study included patients who received cochlear implants at the Auditory Implant Center of the Otorhinolaryngology-Head and Neck Surgery, China PLA General Hospital;
* 2. The patients ranged from 16 to 90 years old;
* 3. The patient experienced hearing loss and had either tinnitus longer than 0.25 years (experimental group 1) or no tinnitus (control group 2) before the cochlear implant surgery;
* 4. The cochlear implants accepted by patients included products from MED-EL, Cochlear, Advanced Bionics and Nurotron;
* 5. All patients voluntarily participated in the study.

Exclusion Criteria:

* 1 Tinnitus types exclude non otogenic tinnitus (including tinnitus caused by hypertension, heart disease, hyperthyroidism, neurasthenia, hyperlipidemia, etc.);
* 2 Contraindications of cochlear implant surgery (refer to the guidelines for cochlear implant 2013 of the Chinese Medical Association);
* 3 Intellectual deficiency

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Electrical stimulation channel number | 1 week after operation
  Stimulating basement membrane with cochlear implant electrode to match tinnitus frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 1 month after operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 2 months after operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 3 months after CI operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 4 months after operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 7 months after operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | 13 months after operation
  frequency. The cochlear implant electrode number is recorded.
Electrical stimulation channel number | over 13 months after operation
  frequency. The cochlear implant electrode number is recorded.
Tinnitus characteristic information questionnaire | Pre-operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 1 week after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 1 month after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 2 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 3 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 4 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 7 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | 13 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus characteristic information questionnaire | over 13 months after operation
  A multifactorial and closed-ended questionnaire was developed by our CI center. The demographics and part of the tinnitus descriptions were recorded in Tinnitus Characteristics questionnaire for CI recipients. The patients' basic information, such as gender, age, aetiology, CI side, CI type, and time of deafness was completed by patients. Tinnitus characteristics information, including localization, duration, and type was collected for correlation analysis.
Tinnitus loudness(CI electrical stimulation intensity) | 1 week after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 1 month after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 2 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 3 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 4 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 7 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | 13 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Tinnitus loudness(CI electrical stimulation intensity) | over 13 months after operation
  The tinnitus loudness was matched by the stimulation current level of cochlear implant electrode, The ultimate electrode stimulation current (IµA) is quantified in µA and the tinnitus loudness is recorded in Qtin (nC, 10-9C) (i.e. Qtin=IµA* tp).
Objective electroencephalography-based assessment(EEG) | Pre-operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 1 week after operation
  The EEG waveforms of CI patients were tested, and the amplitude and latency were recorded.
Objective electroencephalography-based assessment(EEG) | 1 month after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 2 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 3 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 4 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 7 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | 13 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | over 13 months after operation
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Speech perception | Pre-operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | 1 months after operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | 2 month after operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | 4 months after operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | 7 months after operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | 13 months after CI operation
  The patient are tested for speech recognition and the results were recorded as a percentage
Speech perception | over 13 months after CI activation
  The patient are tested for speech recognition and the results were recorded as a percentage

SECONDARY OUTCOMES:
Pure tone test | pre-operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | 1 month after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | 2 months after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | 4 months after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | 7 month after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | 13 month after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Pure tone test | over 13 month after operation
  Evaluation of 250-8000hz hearing effect in patients with hearing loss
Self-Rating Anxiety Scale (SAS) questionnaire | Pre-operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | 1 month after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | 2 months after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | 4 months after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | 7 months after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | 13 months after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.
Self-Rating Anxiety Scale (SAS) questionnaire | over 13 months after operation
  Assessment of patients' mental state （depression, anxiety, insomnia），The result analysis chart of this system shows the standard score. The higher the score, the more serious the symptoms in this regard. Generally speaking, those whose total anxiety score is less than 50 are normal; 50-60 is mild, 61-70 is moderate, and more than 70 is severe anxiety. The number of negative items means the number of items on which the subject did not respond, and the number of positive items means the number of items on which the subject responded. Total rough score: the scores of 20 items are added together, and the demarcation score is 40 points.

CONTACTS AND LOCATIONS:
Overall Officials: Shi m Yang, M.D., Ph.D., Study Director — Chinese PLA General Hospital
Locations (1):
- Qian Wang, Beijing, France, China